CLINICAL TRIAL: NCT07135674
Title: Evaluation of Thermoreversible Avocado-based Gel as an Adjunct to Scaling and Root Planing in Chronic Periodontitis Patients: A Clinical And Microbiological Study
Brief Title: Evaluation of a Herbal Antiseptic Gel as a Supportive Treatment for Teeth Cleaning in Patients With Periodontal Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rungta College of Dental Sciences and Research (Other)
Responsible Party: Principal Investigator, Karthik Krishna M, Principal Investigator, Rungta College of Dental Sciences and Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCDSR/IEC/MDS/2023/D-37
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Periodontal Diseases
Keywords: periodontitis; P. gingivalis; P. intermedia; local drug delivery
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scaling and root planing with subgingival application of placebo gel (Placebo Comparator): scaling and root planing of the entire dentition followed by subgingival application of placebo gel in selected site
  Interventions: Drug: placebo gel
- scaling and root planing with subgingival application of thermoreversible herbal gel (Experimental): scaling and root planing of the entire dentition followed by subgingival application of herbal gel in selected site
  Interventions: Drug: herbal drug

INTERVENTIONS:
Drug: placebo gel — local drug delivery of placebo gel
  Arms: scaling and root planing with subgingival application of placebo gel
Drug: herbal drug — local drug delivery of herbal gel
  Arms: scaling and root planing with subgingival application of thermoreversible herbal gel

SUMMARY:
The goal of this clinical trial is to learn if the herbal gel is more effective as compared to placebo in reducing periodontal inflammation in patients with periodontal disease.

The clinicians shall check various periodontal parameters in the subjects over a scheduled duration.

Participants will be administered the gel once subgingivally and the periodontal parameters shall be recorded before gel delivery then again after 1,3 and 6 months.

Plaque samples were taken at baseline and 6 months

DETAILED DESCRIPTION:
Chronic periodontitis is a prevalent inflammatory condition primarily caused by bacterial plaque biofilm, leading to progressive attachment and bone loss. Scaling and root planing (SRP) is the gold standard for its management. Recently, natural and herbal-based adjuncts have gained attention for their antimicrobial and anti-inflammatory properties. This study aimed to evaluate the clinical and microbiological effectiveness of 4% avocado gel as an adjunct to SRP in the treatment of chronic periodontitis.

A randomized controlled clinical trial was conducted on patients diagnosed with chronic periodontitis. Subjects were divided into two groups: Group I received SRP with subgingival application of placebo gel, and Group II received SRP along with subgingival application of 4% avocado gel. Clinical parameters, including Plaque Index (PI), Papilla Bleeding Index (PBI), Probing Pocket Depth (PPD), and Relative Attachment Level (RAL), were recorded at baseline and after 4th week and 12th week. Microbiological analysis was conducted at recorded at baseline, 4th week,12th week and 24th week to assess the presence of Porphyromonas gingivalis and Prevotella intermedia using culture methods.

ELIGIBILITY:
Inclusion Criteria: 1. Patients with Chronic periodontitis having periodontal pockets (non-adjacent sites) of >5mm

Exclusion Criteria:

* history of any systemic disease, Antibiotic treatment during the 6 months period prior to the study, Pregnant and lactating woman, Periodontal treatment during the previous 3 months, Severe caries or extensive restoration on the objective teeth.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Papilla Bleeding Index | 3 months
Plaque Index | 3 months
Probing Pocket Depth | 3 months
Relative Attachment Level | 3 months

SECONDARY OUTCOMES:
CFUs | 6 months
  Colony Forming Units

CONTACTS AND LOCATIONS:
Locations (1):
- Rungta College of Dental Sciences and Research, Durg, Chhattisgarh, India